CLINICAL TRIAL: NCT05077410
Title: Minimal Invasive TLIF Arthrodesis Using Augmented Reality Navigation for Percutaneous Pedicle Aiming
Acronym: ARSN
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7845
Record Dates: First submitted 2021-09-30; First posted 2021-10-14 (Actual); Last update posted 2021-10-14 (Actual); Status verified 2021-09

CONDITIONS: Arthrosis
Keywords: Arthrosis; Spondylolisthesis; Degenerative spondylolisthesis; Arthrodesis; Osteosynthesis-arthrodesis; Fluoroscopy.; Pedicle screws
MeSH Terms: conditions — Osteoarthritis; Spondylolisthesis; Ankylosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Surgery for degenerative spondylolisthesis requires decompression of the narrow lumbar canal and fixation by osteosynthesis-arthrodesis. Conventional surgery is done through the open route. For 10-15 years, minimally invasive techniques have been established, allowing faster postoperative recovery for the patient. The downside to these techniques is the use of intraoperative fluoroscopy. This is why surgical navigation systems have been developed, allowing safe positioning of implants (pedicle screws). A new process (augmented reality navigation) has been tested in vitro and applied in open surgery. The HUS were the first establishment to apply this new method in minimally invasive surgery in a hybrid room of surgery and interventional radiology.

ELIGIBILITY:
Inclusion criteria:

* Major subject (≥18 years old)
* Subject operated at the HUS between March and December 2019
* Subject with a surgical indication for arthrodesis and decompression of the lumbar canal for degenerative spondylolisthesis L3-L4 or L4-L5
* Subject not having expressed his opposition, after information, to the reuse of his data for the purposes of this research.

Exclusion criteria:

* Subject having expressed opposition to participating in the study
* Subject under guardianship or guardianship
* Subject under safeguard of justice

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Major subject with a surgical indication for arthrodesis and decompression of the lumbar canal for degenerative spondylolisthesis L3-L4 or L4-L5
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2021-10-25 (Estimated); Study Completion 2021-10-25 (Estimated)

PRIMARY OUTCOMES:
Retrospective description of minimally invasive surgery using augmented reality navigation | Files analysed retrospectively from March 01, 2019 to December 31, 2019 will be examined]

CONTACTS AND LOCATIONS:
Overall Officials: Yann Philippe YannPhilippe.CHARLES@chru-strasbourg.fr, MD, PhD, Principal Investigator — Service de Chirurgie du Rachis - Hôpitaux Universitaires de Strasbourg
Locations (1):
- Service de Chirurgie du Rachis - Hôpitaux Universitaires de Strasbourg, Strasbourg, France